CLINICAL TRIAL: NCT02164045
Title: Study to Evaluate the Effect of Food on the Pharmacokinetics of BMS-626529 From an Extended-Release Formulation of BMS-663068 in Healthy Subjects
Brief Title: Study to Evaluate the Effect of Food on the Pharmacokinetics of BMS-626529
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 206283; AI438-042 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-663068- Fasted (Experimental): BMS-663068 tablet twice a day by mouth on specified days
  Interventions: Drug: BMS-663068
- BMS-663068- Fed (Experimental): BMS-663068 tablet twice a day by mouth on specified days
  Interventions: Drug: BMS-663068

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068

SUMMARY:
The current food effect study is being performed to support a Phase 3 study with BMS 663068. Results from this study will inform whether patients in the upcoming Phase 3 study can be given the flexibility to dose BMS-663068 in the fasted state, if so desired.

DETAILED DESCRIPTION:
Primary Purpose: Other: To assess the effect of food on the steady-state exposure of BMS-626529 when administered as BMS 663068 600 mg twice daily (BID) to healthy subjects

Acquired Immune Deficiency Syndrome (AIDS)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical and surgical history, physical examination findings, 12-lead ECG measurements, and clinical laboratory test results
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive
* Males and Females, ages 18 to 50 years, inclusive
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (HCG)) within 24 hours prior to the start of study drug

Exclusion Criteria:

* Any significant acute or chronic medical illness as determined by the investigator
* Current or recent (within 3 months of study drug administration) gastrointestinal disease that could impact upon the absorption of study drug
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal surgery that could impact upon the absorption of study drug
* Inability to tolerate oral medication
* Recent (within 6 months of study drug administration) history of smoking or current smokers
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, electrocardiogram (ECG) or clinical laboratory determinations beyond what is consistent with the target population
* Any of the following on 12-lead ECG prior to study drug administration, confirmed by repeat:

  * PR ≥ 210 msec
  * QRS ≥ 120 msec
  * QT ≥ 500 msec
  * QTcF ≥ 450 msec
  * Positive urine screen for drugs of abuse
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or Human Immunodeficiency Virus-1 (HIV-1), -2 antibodies, and HIV-1 RNA

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2014-07-25 (Actual); Study Completion 2014-07-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) for BMS-626529 in the presence and absence of food | Days 1-4 of Periods 1 and 2
Area under the concentration-time curve in one dosing interval (AUC(TAU)) for BMS-626529 in the presence and absence of food | Days 1-4 of Periods 1 and 2

SECONDARY OUTCOMES:
Safety and tolerability endpoints including incidence of Adverse events (AEs), serious AEs, AEs leading to discontinuations, deaths, and the results of vital signs, ECGs, physical examinations, and clinical laboratory tests | Approximately up to 41 days
Time of maximum observed plasma concentration (Tmax) of BMS-626529 | Day 4 of each period
Plasma concentration observed at 12 hours postdose (C12) of BMS-626529 | Day 4 of each period
Trough observed plasma concentration (Ctrough) of BMS-626529 | Days 1-4 of each period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, San Antonio, Texas, United States